CLINICAL TRIAL: NCT04045704
Title: The Effects of Unilateral and Bilateral Cataract Extraction on Visual Function of Advanced Age-Related Macular Degeneration Patients.
Brief Title: Cataract Surgery on Advanced Age Related Macular Degeneration Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No study coordinator available. No patient recruitment possible.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jeffrey Chambers, Clinical Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19-00830
Record Dates: First submitted 2019-07-17; First posted 2019-08-05 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Cataract; Macular Degeneration Advanced
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cataract Surgery — Patients with bilateral Advanced Age-related macular degeneration and concurrent cataracts will be receiving bilateral cataract surgery

SUMMARY:
The degree at which cataract surgery improves visual function in patients with advanced age-related macular degeneration (Advanced AMD) has been an on-going topic of discussion. Our objective in this study is to determine if patients with Advanced AMD and concurrent cataracts will experience greater improvement in their quality of life from having cataract surgery on one or both eyes. The findings from this project will provide evidence for clinical decision making on whether performing bilateral cataract surgery on Advanced AMD patients is cost-effective and worth the second surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients above the age of fifty with both Advanced AMD and Cataracts bilaterally from the Okanagan Valley will be selected for this study.

Patients who chose to have bilateral cataract surgery, were able to understand the research parameters, and had no other severe eye disease that may distort the studies results.

Patients will be selected for the study according to the National Eye Institute definition of Advanced AMD.

"Advanced AMD (AREDS category 4) is characterized by one or more of the following (in the absence of other causes) in one eye:

Geographic atrophy of the RPE involving the foveal center.

Neovascular maculopathy that includes the following:

* Choroidal neovascularization (CNV) defined as pathologic angiogenesis originating from the choroidal vasculature that extends through a defect in Bruch's membrane
* Serous and/or hemorrhagic detachment of the neurosensory retina or RPE
* Retinal hard exudates (a secondary phenomenon resulting from chronic intravascular leakage)
* Subretinal and sub-RPE fibrovascular proliferation
* Disciform scar (subretinal fibrosis)"

Exclusion Criteria:

* Severe intraoperative or postoperative complications such as retinal detachments, and capsule ruptures
* Inability to complete the required testing (auto-refractive and visual acuity)
* Inability to attend appointments
* Inability to complete the questionnaire with Co-I assistance
* Severe eye disease that may distort the studies results such as but not limited to Epithelial Basement Membrane Dystrophy (EBMD) and retinal detachments.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Life style Questionnaire to determine change in visual function. | Through study completion, an average of 1 year
  Our primary outcome will be a life style questionnaire (qualitative) to determine the change in visual function from baseline to after surgery.
  This questionnaire includes 25 close-ended questions that are graded on a 5 point grading scale from 1 (great difficulty due to vision) and 5 (no problem due to vision). The questions can also be graded as not applicable to an individuals life, or 0 being something there are no longer possible to do, due to vision.
  The 25 close-ended questions are divided into 4 sub-scales:
  1. Distance Vision, Mobility, and Lighting (Q: 1-12)
  2. Adjustment (Q:13-16)
  3. Reading and Fine Work (Q: 17-21)
  4. Activities of Daily Living (Q: 22-25)
  A total score can range from a 125 indicating best visual function to 0 indicating complete loss of visual function.

SECONDARY OUTCOMES:
Snellens Chart to determine change in visual acuity | Through study completion, an average of 1 year
  Quantitative measure of a patients visual acuity. Change from baseline visual acuity to after surgery on both eyes.
Auto Refractive to determine change in visual acuity | Through study completion, an average of 1 year
  An auto-refractor is a computerized machine to measure patients visual acuity. Change from baseline visual acuity to after surgery on both eyes.

IPD SHARING:
Plan to Share IPD: Undecided